CLINICAL TRIAL: NCT02898545
Title: Recurrent Atrial Fibrillation
Acronym: Recurrent AF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Cincinnati (Other)
Responsible Party: Principal Investigator, Mehran Attari, Principal Investigator, University of Cincinnati
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 2015-2478
Record Dates: First submitted 2016-09-08; First posted 2016-09-13 (Estimated); Last update posted 2017-08-01 (Actual); Status verified 2017-07

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- SEEQ monitor (Other): Subjects will be monitored via use of the SEEQ monitor
  Interventions: Device: SEEQ monitor
- Standard of care (No Intervention): Subjects will not wear the SEEQ monitor or may have a pre-existing implanted device capable of detecting atrial fibrillation

INTERVENTIONS:
Device: SEEQ monitor — An external cardiac rhythm monitor
  Arms: SEEQ monitor

SUMMARY:
This study will evaluate the recurrence rates of atrial fibrillation that develops in the hospital following non cardiac procedures or surgeries or acute medical illnesses.

DETAILED DESCRIPTION:
Eligible individuals with no previous history of atrial fibrillation or flutter who develop a limited episode of atrial fibrillation during a hospital stay for an acute medical illness or non-cardiothoracic surgery or procedure. Patients will be monitored for a period of 1 month using Medtronic SEEQ monitors for recurrence. Subjects will self assign to wear the SEEQ monitor or standard of care. Individuals with implanted cardiac devices capable of detecting atrial fibrillation will also be included.

ELIGIBILITY:
Inclusion Criteria:

* Development of atrial fibrillation or flutter during a hospital stay following a non-cardiac procedure or acute medical illness
* CHADS2VASc score of 2 or more

Exclusion Criteria:

* Prior history of atrial fibrillation of flutter
* Requiring ventilator support or in shock
* Acute decompensated heart failure or EF =/< 40%
* Greater than mild valvular heart disease
* Other structural heart disease such as more than mild LVH, constrictive or restrictive cardiomyopathy
* Hyperthyroidism uncontrolled at the time of diagnosis if known
* Pulmonary embolism that requires thrombolysis or resulted in shock
* Use of antiarrhythmic drugs (class I or III) at the time of discharge
* Cardiothoracic surgery in the last 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2016-09; Primary Completion 2017-07-20 (Actual); Study Completion 2017-07-20 (Actual)

PRIMARY OUTCOMES:
Recurrence of atrial fibrillation | 28 days
  The rate of recurrence of atrial fibrillation will be compared to the recurrence noted in the standard of care arm.

CONTACTS AND LOCATIONS:
Overall Officials: Mehran Attari, MD, Principal Investigator — University of Cincinnati
Locations (1):
- University of Cincinnati Medical Center, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: Undecided